CLINICAL TRIAL: NCT04999618
Title: DOUBLE-SKIN: a New Approach in Laser Surgery Using the Regenerative Solution in Children Diagnosed With Vascular Pathology: a Randomised, Double-blind, Placebo-controlled Trial
Brief Title: A New Approach in Laser Surgery Using the Regenerative Solution in Children Diagnosed With Vascular Pathology
Acronym: DOUBLE-SKIN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Center for Vascular Pathology, Moscow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CVPMoscow
Record Dates: First submitted 2021-07-17; First posted 2021-08-11 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Vascular Diseases; Vascular Malformation; Capillary Malformation-Arteriovenous Malformation; Port-Wine Stain; Sturge-Weber Syndrome; Vascular Tumor
Keywords: Vascular Diseases; Laser treatment; Capillary Malformation; Port-Wine Stain; Vascular Tumor
MeSH Terms: conditions — Vascular Diseases; Vascular Malformations; Capillary Malformation-Arteriovenous Malformation; Port-Wine Stain; Sturge-Weber Syndrome; Vascular Neoplasms; Capillary Malformations, Congenital, 1

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, clinicians and the research team, completing baseline and follow-up assessments were masked to group allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group with Haemoblock (A) (Active Comparator)
  Interventions: Drug: Haemoblock
- Group without Haemoblock (B) (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Haemoblock — Delivering with transdermal patches
  Arms: Group with Haemoblock (A)
Other: Placebo — Delivering with transdermal patches
  Arms: Group without Haemoblock (B)

SUMMARY:
Laser treatment (LT) is the first-line treatment for Vascular Pathology. However even when LT is based on the selective photothermolysis it causes the first-degree burns. While being typically benign by affecting only the epidermis, or outer layer of skin, the burn site is remaining red, dry, and very painful. As Haemoblock contains nanoparticles of silver and is known for both bactericidal and bacteriostatic effects, it likely decreases the potential for infection postoperatively. Furthermore, after fibrin replaces the superficial structure "Hemoblock-albumin", the polyacrylate matrix is plasmolyzed which initiates the cascade of signals required for the tissue regeneration processes. Objective of the study was to examine the effect of the Regenerative Solution "Hemoblock" in lowering postoperative complications in children diagnosed with Vascular Pathology undergoing a laser surgery if delivered with transdermal patches.

ELIGIBILITY:
Inclusion Criteria:

* clinically diagnosed Vascular Pathology

Exclusion Criteria:

* age
* severe allergic reaction

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2021-10-27 (Actual)

PRIMARY OUTCOMES:
Preventing negative outcomes of postoperative infection | Early postoperative period and at 3 weeks
  Validated scales

SECONDARY OUTCOMES:
Preventing prolonged functional recovery | Early postoperative period and at 3 weeks
  Validated scales

OTHER OUTCOMES:
Preventing likelihood of mental health issues | Early postoperative period and at 3 weeks
  Validated scales

CONTACTS AND LOCATIONS:
Overall Officials: Ekaterina M Listovskaya, BSc, Principal Investigator — The Vascular Anomalies Center (VAC) "Hemangioma",; Dmitry V Romanov, MD, Study Chair — The Vascular Anomalies Center (VAC) "Hemangioma"; Alexander Plotkin, PhD, Study Chair — Moscow Regional Research Institute of Blood
Locations (1):
- The Vascular Anomalies Center (VAC) "Hemangioma", Moscow, Russia